CLINICAL TRIAL: NCT07251777
Title: Prone vs Supine Position in Potential Organ Donors: PRODONAR Multicenter Clinical Trial
Brief Title: Prone vs Supine Position in Potential Organ Donors: Multicenter Clinical Trial
Acronym: PRODONAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Alta Complejidad del Bicentenario Esteban Echeverría (Other Government)
Collaborators: Hospital Cuenca Alta Néstor Kirchner Cañuelas (Unknown); Hospital Escuela General José Francisco de San Martín (Corrientes) (Unknown); Hospital Ángel Cruz Padilla (Tucuman) (Unknown); Hospital Central de Mendoza (Unknown); Hospital Simplemente Evita de Gonzalez Catan (Unknown); HIGA Abraham Piñeyro (Unknown); Hospital San Martín (Entre Ríos) (Unknown); Hospital Interzonal General de Agudos San Roque (Unknown); Hospital Regional Dr. Enrique Vera Barros (La Rioja) (Unknown); Instituto Nacional Central Único Coordinador de Ablación e Implante (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1168576558
Record Dates: First submitted 2024-01-26; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Prone Position; Donors; Lung Procurement; Tissue Donors; Lung Transplantation
Keywords: Prone position; Donors; Lung procurement; Tissue donors; Mechanical Ventilation; Brain Death; Lung Transplantation
MeSH Terms: conditions — Brain Death | interventions — Prone Position

STUDY DESIGN:
Intervention Model Description: The PRODON-AR study is a prospective, longitudinal, multicenter, randomized, parallel group, unblinded trial with electronic-based randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prone position (Experimental): Potential donors assigned to the experimental group will be placed in a prone position. This position will be maintained until one hour prior to entering the operating room for organ ablation.
  Interventions: Procedure: Prone position
- Supine position (No Intervention): Potential donors assigned to the control group (supine position) will continue in that position with the usual treatment.

INTERVENTIONS:
Procedure: Prone position — The only intervention that differs between the groups will be that the potential donors assigned to the experimental group will be kept in a prone position until they enter the operating room for ablation.
  Arms: Prone position

SUMMARY:
Background and justification: In Argentina, 9,650 people are on the organ transplant waiting list, including 290 who require a lung transplant. In 2022, 21 unilateral lungs, 18 bilateral lungs, and one cardiopulmonary block were implanted, representing only 1.9% of all transplants. Maintaining organ viability in potential donors (PD) is challenging because brain death triggers adrenergic activation, hemodynamic instability, and atelectasis due to mechanical ventilation and loss of respiratory muscle activity. These factors impair gas exchange and reduce the number of lungs suitable for transplantation.

Ventilatory management in PDs aims to preserve lung function, minimize risks of invasive mechanical ventilation (IMV), and maintain adequate gas exchange while preventing alveolar collapse and overdistension. Strategies derived from Acute Respiratory Distress Syndrome (ARDS) include recruitment maneuvers, which may cause complications. In contrast, prone positioning improves ventilation-perfusion matching and increases functional lung parenchyma.

This study proposes prone positioning as a preventive ventilatory strategy to optimize lung preservation in organ donors.

Objectives: (1) Determine whether early prone positioning after BD certification increases the proportion of lungs meeting suitability criteria for transplantation. (2) Evaluate its effect on the availability of other transplantable organs and on hemodynamic stability.

Methods: The PRODON-AR study is a prospective, multicenter, randomized controlled trial conducted in 10 intensive care units (ICUs) across Argentina. Recruitment began on June 1, 2023, and will continue until 250 PDs are enrolled. Participants will be randomly assigned to standard care (supine) or prone positioning following BD certification. Eligible donors will be those with confirmed BD, meeting multi-organ donation criteria, and without documented opposition to donation. Exclusion criteria include contraindications to prone positioning. Donors will be excluded from analysis if the interval between BD certification and proning exceeds 12 hours, if more than 20% of data for key variables are missing, or if clinical conditions require returning to the supine position.

The primary outcome is the number of lungs suitable for transplantation. Secondary outcomes include the number of organs transplanted, vasopressor requirements, and variables related to gas exchange and respiratory mechanics.

DETAILED DESCRIPTION:
This protocol follows the SPIRIT guidelines (Standard Protocol Items: Recommendations for Interventional Trials).

Introduction: Organ transplantation replaces a failing organ with one from a donor. Ablation enables organ removal for therapeutic use in recipients with terminal organ failure. In Argentina, as of February 2023, 9,650 people were on the national waiting list, including 290 requiring lung transplantation. In 2022, 767 real donors generated 2,090 organs, of which only 40 lungs were transplanted, representing 1.9% of all transplants.

The lung remains one of the most challenging organs for procurement due to strict selection criteria and rapid functional deterioration after brain death (BD). Countries such as Spain, which lead global donation rates, have broadened donor criteria ("expanded criteria donors"), demonstrating that the use of marginal lungs does not increase recipient mortality.

Following BD, sympathetic nervous system activation triggers a massive inflammatory response leading to endothelial and alveolar damage. Potential donors (PDs) under invasive mechanical ventilation (IMV) experience additional inflammatory stress. Neuromuscular paralysis and a lack of respiratory effort promote atelectasis, particularly in dependent lung regions, thereby compromising ventilation-perfusion (V/Q) matching. The apnea test and FiO₂ 100% exposure can worsen atelectasis through nitrogen washout. In addition, an absent cough reflex predisposes to secretion retention and infection, reducing lung viability and secondarily impairing the function of other organs through systemic hypoxia and inflammation.

Rationale: Ventilatory management in PDs aims to preserve lung function, reduce IMV-induced injury, and maintain optimal gas exchange while preventing alveolar collapse and overdistension. Lung-protective ventilation (tidal volume 6-8 mL/kg predicted body weight and adequate positive end-expiratory pressure, PEEP) remains standard; however, the proportion of suitable lungs for procurement remains low.

Recruitment maneuvers, formerly used in ARDS, are now avoided due to their association with increased mortality (ART trial, 2018). In turn, prone positioning (PP) has proven several clinical benefits in ARDS, enhancing oxygenation and reducing ventilator-induced lung injury. PP promotes more homogeneous ventilation, recruits dorsal lung areas, enhances oxygenation, and improves right ventricular function without significant hemodynamic compromise. Studies such as PROSEVA demonstrated reduced cardiac arrests and better extrapulmonary organ function in PP patients.

In PDs, PP could similarly improve oxygenation and hemodynamics, facilitating donor management and increasing organ suitability. The PRODON-AR study will test whether PP after BD certification increases the proportion of lungs suitable for transplantation compared with standard supine positioning (SP).

Primary objective: Evaluate whether early PP after BD certification increases the number of lungs meeting suitability criteria for transplantation. Secondary objective: Assess the effect of PP on hemodynamic stability and on the availability of other transplantable organs.

Methods

Design: The PRODON-AR study is a prospective, multicenter, randomized controlled trial (RCT) conducted across 11 intensive care units (ICUs) in Argentina. Recruitment began on June 1, 2023, and will continue until 250 PDs are enrolled. Participants will be randomized to PP (intervention) or SP (control). Randomization will be electronic and unblinded.

Inclusion criteria: confirmed BD according to national protocol, eligibility for multi-organ donation, and no documented opposition to donation.

Exclusion criteria: contraindications to PP (e.g., spinal instability, major abdominal wounds). PDs will be excluded from analysis if the interval between BD certification and PP exceeds 12 h, more than 20% of key variable data are missing, or if medical conditions require return to SP.

Procedure: After BD certification, ventilation will be set in VC-CMV mode with tidal volume 6-8 mL/kg predicted body weight, PEEP 8-12 cmH₂O, respiratory rate to maintain PaCO₂ 35-45 mmHg, FiO₂ for SpO₂ 94-98%, and inspiratory time 0.8-1.0 s.

Baseline evaluation (in SP) includes:

* Chest X-ray or CT for infiltrates,
* Respiratory mechanics (peak, plateau, total PEEP, ΔP, compliance, resistance),
* Optional lung ultrasound for aeration scoring,
* Arterial blood gas (PaO₂/FiO₂, base excess, bicarbonate, SpO₂),
* Vasopressor requirement (μg/kg/min),
* Intra-abdominal pressure (mmHg) and urine output (mL/h).

After baseline, PDs will be randomized to PP or SP. Those assigned to PP will be turned following institutional protocols. Reassessment will occur 8-12 h after randomization and again before organ procurement. Complications will be recorded. In the PP group, the donor remains prone until preparation for surgery, with head and limb repositioning every 3 h. For procurement, all donors are returned to SP before transfer to the operating room.

Outcomes Primary: number of lungs suitable for transplantation. Secondary: number of organs transplanted, PaO₂/FiO₂ ratio, respiratory mechanics, vasopressor requirement, and hemodynamic variables.

Statistical Analysis Descriptive statistics (mean, median, SD, IQR) will summarize continuous variables. Categorical variables will be expressed as frequencies and percentages.

Inferential analysis:

Primary outcome: logistic regression assessing the association between PP and lung suitability, adjusted for age, sex, time from BD to PP, and comorbidities (odds ratio with 95% CI).

Secondary outcomes: group comparisons via t-test/ANOVA or Mann-Whitney/Kruskal-Wallis as appropriate. P<0.05 will indicate significance. Subgroup analysis will explore the effect of PP timing and presence of atelectasis. Analyses will use JASP (version 2021).

Sample Size: Based on a 6% baseline lung suitability rate (per INCUCAI data), 10% expected improvement, α=0.05, power=80%, and 10% anticipated loss, a total of 250 PDs (125/group) will be required using Student's t-test for proportions.

Ethics: The trial addresses the critical shortage of transplantable lungs in Argentina. Evidence for PP benefits in critical care is robust, yet data in PDs after BD remain scarce. The study involves deceased individuals with certified BD under national law (Laws 17.132, 25.326, 26.629, 27.447, and Decree 1089/2012), posing no risk to living persons. In turn, this study was officially reviewed and approved by the Ministry of Health of Argentina, managed by the research ethics committee (REC) of INCUCAI (INSTITUTO NACIONAL CENTRAL ÚNICO COORDINADOR DE ABLACIÓN E IMPLANTE), under the reference number EX-2024-43540732-APN-INCUCAI#MS.

All data will be anonymized per data protection regulations. Inclusion of deceased donors does not require informed consent (Law 27.447, Chapter VIII; CIOMS Guideline 10 exception). The study does not interfere with organ procurement and relies on standard clinical measurements already documented in SINTRA (National Information System for Procurement and Transplantation).

Biological samples are limited to routine blood and urine analyses and discarded immediately after testing. No genetic studies or material storage are planned. Each site is led by an experienced transplant professional. The principal investigator has extensive experience in donor management and research coordination.

Confidentiality: All participant data will remain confidential. Only anonymized and authorized information will be used for analysis and publication.

Results Publication Policy: Findings will be submitted to high-impact journals and shared with the Argentine Societies of Medicine, Intensive Care, and Transplantation. Ethical and legal publication standards, including conflict-of-interest disclosure, will be strictly followed.

Conflict of Interest: The investigators declare no conflicts of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patients who died under neurological criteria
* 18 to 70 years of age
* Meet multi-organ donor criteria
* That they have no opposition to the donation.

Exclusion Criteria:

* Patients who have expressly stated that they do not donate organs
* Patients who, for some reason, cannot establish a prone position
* Deceased with contraindication for organ donation.

Elimination criteria

* Time between diagnosis of ME and prone greater than 12 hours
* Loss of more than 20% of data on main variables.
* Require changing a patient from the prone to the supine position for any reason

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Potential lung donor | The assessment will be conducted within 1 hour before the potential donor enters the operating room for organ ablation.
  Before the potential donor enters the operating room for organ ablation, it will be determined whether the individual is eligible to be a lung donor based on the criteria established by the Spanish Transplant Society

SECONDARY OUTCOMES:
Organs ablated and implanted | Data will be collected from the INCUCAI website up to 2 days post-ablation, following the procedure
  The organs ablated from each subject will be recorded, as well as which of them were actually implanted in a recipient.
Vasopressor requirement | The vasopressor requirement will be evaluated at three time points: 1. Immediately after the diagnosis of brain death (BD) 2. At 12 hours after the diagnosis of BD 3. Prior to entering the operating room for organ ablation
  The requirement for vasopressor drugs will be recorded, including the specific drug(s) used and the dose administered, expressed in mcg/kg/min.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Centeno, Dr., Principal Investigator — Hospital de Alta Complejidad del Bicentenario Esteban Echeverría
Locations (1):
- Hospital de Alta Complejidad del Bicentenario Esteban Echeverría, Monte Grande, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Maciel CB, Greer DM. ICU Management of the Potential Organ Donor: State of the Art. Curr Neurol Neurosci Rep. 2016 Sep;16(9):86. doi: 10.1007/s11910-016-0682-1. PMID 27498101
- [Background] Del Rio F, Escudero D, De La Calle B, Vidal FG, Paredes MV, Nunez JR. [Evaluation and maintenance of the lung donor]. Med Intensiva. 2009 Jan-Feb;33(1):40-9. doi: 10.1016/s0210-5691(09)70304-3. Spanish. PMID 19232208
- [Background] Meyfroidt G, Gunst J, Martin-Loeches I, Smith M, Robba C, Taccone FS, Citerio G. Management of the brain-dead donor in the ICU: general and specific therapy to improve transplantable organ quality. Intensive Care Med. 2019 Mar;45(3):343-353. doi: 10.1007/s00134-019-05551-y. Epub 2019 Feb 11. PMID 30741327
- [Background] Bansal R, Esan A, Hess D, Angel LF, Levine SM, George T, Raoof S. Mechanical ventilatory support in potential lung donor patients. Chest. 2014 Jul;146(1):220-227. doi: 10.1378/chest.12-2745. PMID 25010965
- [Background] Writing Group for the Alveolar Recruitment for Acute Respiratory Distress Syndrome Trial (ART) Investigators; Cavalcanti AB, Suzumura EA, Laranjeira LN, Paisani DM, Damiani LP, Guimaraes HP, Romano ER, Regenga MM, Taniguchi LNT, Teixeira C, Pinheiro de Oliveira R, Machado FR, Diaz-Quijano FA, Filho MSA, Maia IS, Caser EB, Filho WO, Borges MC, Martins PA, Matsui M, Ospina-Tascon GA, Giancursi TS, Giraldo-Ramirez ND, Vieira SRR, Assef MDGPL, Hasan MS, Szczeklik W, Rios F, Amato MBP, Berwanger O, Ribeiro de Carvalho CR. Effect of Lung Recruitment and Titrated Positive End-Expiratory Pressure (PEEP) vs Low PEEP on Mortality in Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2017 Oct 10;318(14):1335-1345. doi: 10.1001/jama.2017.14171. PMID 28973363
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Vieillard-Baron A, Charron C, Caille V, Belliard G, Page B, Jardin F. Prone positioning unloads the right ventricle in severe ARDS. Chest. 2007 Nov;132(5):1440-6. doi: 10.1378/chest.07-1013. Epub 2007 Oct 9. PMID 17925425
- [Background] Matejovic M, Rokyta R Jr, Radermacher P, Krouzecky A, Sramek V, Novak I. Effect of prone position on hepato-splanchnic hemodynamics in acute lung injury. Intensive Care Med. 2002 Dec;28(12):1750-5. doi: 10.1007/s00134-002-1524-y. Epub 2002 Oct 26. PMID 12447518
- See also: Ministerio de Salud de Argentina — https://www.argentina.gob.ar/sites/default/files/resolucion_716_2019_anexo_i.pdf
- See also: It is the computer system for the administration, management, supervision and consultation of the procurement and transplantation of organs, tissues and cells at the national level. — https://sintra.incucai.gov.ar/